CLINICAL TRIAL: NCT03021798
Title: Characterising SARcopenia and Sarcopenic Obesity in Patients Aged 65 Years and Over at Risk of Mobility Disability. An OBServational Clinical Trial (SARA-OBS)
Brief Title: An OBServational Clinical Trial (SARA-OBS) in Sarcopenia and Sarcopenic Obesity in Patients Aged 65 Years and Over
Acronym: SARA-OBS
Status: Completed | Type: Observational
Sponsor: Biophytis (Industry)
Responsible Party: Sponsor
Other Study IDs: BIO101-CL02
Record Dates: First submitted 2017-01-03; First posted 2017-01-16 (Estimated); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Sarcopenia; Gait Disorders in Old Age; Muscle Weakness
Keywords: Sarcopenia; Sarcopenic Obesity; observational study; 6-minute walking distance; 400 meters walking test; Patient Reported Outcomes
MeSH Terms: conditions — Sarcopenia; Muscle Weakness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No Drug and no aspecific intervention — No intervention

SUMMARY:
The SARA-OBS is a single arm phase 2 clinical trial, with no investigational product and no therapeutic intervention that will be conducted in three European countries, (Belgium, France and Italy), and in the US.

300 community dwelling older adults (men or women≥65 years) reporting loss of physical function and at risk of mobility disability, will undergo mobility functional evaluation and Dual-energy X-ray Absorptiometry DXA scan for body composition determination twice, at six-month interval.

Participants aged ≥ 65 years complaining of poor physical function will be selected to perform SPPB (Short Physical Performance Battery)tests. Those with SPPB scores ≤ 8/12 will be selected to perform body composition analysis with DXA Scan. Participants with ALM/BMI < 0.789 in men and 0.512 in women will be included. The investigational phase will comprise two main visits: the inclusion visit and the 6-month visit. Both the 6-minute walk distance test and the 400-metre walking test will be administered at the main visits. Patient Reported Outcomes (PROs) will be completed by the patients at the same visits.

DETAILED DESCRIPTION:
The SARA-OBS is a phase 2 clinical trial, with no investigational product and no therapeutic intervention. It will be conducted in three European countries, Belgium, France and Italy, and in the US.

300 community dwelling older adults (men or women≥65 years) reporting loss of physical function and at risk of mobility disability, will undergo mobility functional evaluation and Dual-energy X-ray Absorptiometry DXA scan for body composition determination twice, at six-month interval.

The general objective is to characterise sarcopenia including "sarcopenic obesity" in a population of older persons living in the community and at risk of mobility disability; evaluate their physical performance and body composition in view of the design of a phase 2 clinical study on the efficacy and safety of BIO101 on the prevention of mobility disability in the at-risk community dwelling older adults (≥65 years) reporting loss of physical function.

The primary objective characterise sarcopenia including sarcopenic obesity, in older persons at risk of mobility disability. Sarcopenia will be defined according to the criteria of the Foundation of NIH; the risk of mobility disability will be operationalised by the Short Physical Performance Battery (SPPB). For this purpose, the 6-minute walking distance and the 400-meter walking test will be evaluated at 6-month intervals, in the absence of any therapeutic intervention. The incident rate of change will be estimated on the sample and pre-specified subgroups (e.g. gender, SPPB baseline score, etc.).

Two important Secondary Objectives are also included :

1. To evaluate muscle strength (handgrip/knee extension) and stair power climbing test
2. To evaluate self-administered quality-of-life tests as putative patient reported outcomes (PROs): Short Form Health Survey (SF-36) and Sarcopenia Quality of Life (SarQol) for all subjects; in addition, TSD-OC for participants with BMI≥30

Exploratory objectives are :

1. To measure tentative biomarkers of sarcopenia and poor physical performance, and test their correlation with physical function change over the study observation.
2. To record actimetry via a connected wearable device, in order to describe daily physical activity and possibly identify patterns predictive of improvement/worsening of physical function.

Primary endpoints are the 6-minute Walk Test/400m Walking Test and Co-Primary endpoints are SF-36 and SarQoL for all subjects; additionally TSD-OC for subjects with BMI ≥ 30.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged ≥ 65 years and living in the community, reporting loss of physical function
2. Short Physical Performance Battery (SPPB) score ≤ 8
3. ALM/BMI < 0.789 in men and 0.512 in women, by DXA scan

Exclusion Criteria:

1. Unable or unwilling to provide informed consent
2. Unable to understand and perform the functional tests, as judged by the Investigator
3. Current treatment with anabolic drugs, i.e. testosterone
4. Clinical conditions:

   1. Current diagnosis major psychiatric disorders.
   2. Alcohol abuse or dependence
   3. Severe arthritis
   4. Cancer requiring active treatment
   5. Lung disease requiring regular use of supplemental oxygen
   6. Inflammatory conditions requiring regular use of oral or parenteral corticosteroid agents
   7. Severe cardiovascular disease (including New York Heart Association [NYHA] class III or IV congestive heart failure, clinically significant valvular disease, history of cardiac arrest, presence of an implantable defibrillator, or uncontrolled angina)
   8. Parkinson's disease or other progressive neurological disorder
   9. Renal disease requiring dialysis
   10. Chest pain, severe shortness of breath, or occurrence of other safety concerns during the baseline the 6MWT, or the 400-meter walk test
5. Current physical/rehabilitation therapy
6. Current enrolment in another clinical trial
7. Concomitant condition implying life expectancy ≤ 6 months
8. Any other condition precluding the regular participation to the clinical trial, as judged by the Investigator.

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: 300 community dwelling older adults (men or women≥65 years) reporting loss of physical function and at risk of mobility disability
Sampling Method: Probability Sample
Enrollment: 218 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
6-minute or 400 meters walk. | Change from Baseline 6 minute or 400 meters to measurement at 6 months.
  The 6 minutes walking distance is a functional exercise capacity test that involves measuring the distance covered by a participant within a specified time of 6 minutes. The 400 meter walking test is a measure of how long it will take for a volunteer to complete the specified 400 meters distance.

SECONDARY OUTCOMES:
SPPB | Change from Baseline SPPB to measurement at 6 months.
  Physical performance tests corresponding to standing balance, walking speed and chair stand will be assessed
DEXA | Change from Baseline DEXA to measurement at 6 months.
  Body composition especially Lean Body Mass and Fat Mass will be measured. This will allow definition of the appendicular Lean Body mass.
Stair Climb Power Test | Change from Baseline Stair Climb Power Test to measurement at 6 months.
  The ability to ascend and descend stairs (9 stairs of 20 cm height) will be assessed in a specific period of time
Actimetry | Change from actimetry at Month1 to measurement at 6 months.
  The continuous physical activity of the volunteers will be recorded using a specific device during the 6-month study period.
Grip strength | Change from Baseline Grip Strength to measurement at 6 months.
  The grip strength will be measured using the appropriate dynamometer. Strength will be measured 3 times for both hands and the highest value will be kept for further analysis.
Knee extension | Change from Baseline knee extension to measurement at 6 months.
  The knee extension measurement will be performed using isokinetic dynamometer.
Patient Reported Outcome : SF-36 | Change from Baseline Patient Reported Outcome to measurement at 6 months.
  Electronically self administrated Patient Reported Outcome SF-36 will be assessed a SF-36 questionnaire.
Patient Reported Outcomes : SarQoL | Change from Baseline Patient Reported Outcome to measurement at 6 months.
  Electronically self administrated Patient Reported Outcome SarQoL will be assessed through the SarQoL questionnaire.
Patient Reported Outcomes TSC-OD for patients with BMI>30 | Change from Baseline Patient Reported Outcome to measurement at 6 months.
  Electronically self administrated Patient Reported Outcomes will be assessed through the TSD-OC questionnaire for volunteers having BMI>30
Patient Reported Outcomes (PAT-D) | Change from Baseline Patient Reported Outcome to measurement at 6 months.
  Electronically administrated Patient Reported Outcome will be assessed with assistance of the investigator through the PAT-D questionnaire.
Biomarkers | Change from Baseline Biomarkers to measurement at 6 months
  Biomarkers specific to Sarcopenia and to the Renin Angiotensin System ( Aldosterone; Renin; Myostatin; PIIINP; IL-6; hsCRP etc....) will be measured at baseline and at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Agus, MD, Study Director — Biophytis
Locations (7):
- United States (3):
  - Institut On Aging, Gainesville, Florida
  - Jean Mayer USDA Human Nutrition research Center on Aging Tufts University, Boston, Massachusetts
  - Columbia University New York, New York, New York
- Université de Liège, Liège, Belgium
- France (2):
  - Centre Hospitalier Lyon Sud 165 Chemin du Grand Revoyet, Pierre-Bénite
  - Gérontopole Toulouse, Toulouse
- Sapienza University of Rome, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fielding RA, Rolland Y, Bruyere O, Desvarieux M, Donini LM, Incalzi RA, Muscaritoli M, Tchalla A, Bonnefoy M, Rondanelli M, Van Maanen R, Mariani J, Margalef C, Del Signore S, Tourette C, Dioh W, Veillet S. Characterizing sarcopenia and sarcopenic obesity in patients aged 65 years and over, at risk of mobility disability: a multicenter observational trial (SARA-OBS). BMC Geriatr. 2025 Aug 4;25(1):590. doi: 10.1186/s12877-025-05895-9. PMID 40759914